CLINICAL TRIAL: NCT02692664
Title: Prospective Multicenter Study for the Endovascular Treatment of Iliac Aneurysm With the Branched E-liac Stent Graft
Acronym: TAILOR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TAILOR
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Iliac Aneurysm; AAA
Keywords: iliac side branch
MeSH Terms: conditions — Iliac Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endovascular aorto-iliac repair
  Other Names: EVAR

SUMMARY:
In this study, patients will be observed who receive an E-liac Stent Graft for treatment of isolated iliac aneurysms or an E-liac Stent Graft in combination with one of the following AAA stent grafts: E-tegra Stent Graft, Endurant AAA Stent Graft, Zenith AAA Endovascular Graft, Gore Excluder AAA Endoprosthesis for treatment of aorto-iliac aneurysms.

Objectives of this post-market registry are:

Primary: To prevent the risk of rupture and death by the treatment of common iliac aneurysm with an iliac branched stent graft (E-liac, JOTEC) Secondary: Evaluation of safety and feasibility of the E-liac Stent Graft System used in endovascular treatment of uni- or bilateral aorto-iliac or iliac aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral aorto-iliac or iliac aneurysm
* Suitable for endovascular repair
* Patient must be compliant with life- long follow-up investigations
* >18 years old
* lliac/femoral access vessel morphology compatible with the implantation procedure and the 18Fr (6mm OD) delivery system
* Non-aneurysmal common iliac artery landing area in case of iliac artery aneurysm ≥ 20mm
* Diameter of the common iliac artery in the proximal landing area: 12mm to 17mm
* Non-aneurysmal external iliac artery segment distal to the aneurysm ≥15mm
* Diameter of the external iliac artery in the distal landing area: 8mm to 13mm
* Non-aneurysmal internal iliac artery segment distal to the aneurysm ≥15mm
* Angle between external iliac artery and internal iliac artery ≤50°
* Thrombus free iliac lumen in the area of iliac bifurcation to open hypogastric side branch and to implant covered stent ≥18mm
* Sufficiently open internal iliac arterv ostium
* Patients must comply with the instructions for use.
* Patients with common iliac aneurysm with a diameter ≥30mm when isolated or common iliac aneurysm with a diameter >25mm when associated with an abdominal aortic aneurysm
* Unilateral or bilateral common iliac aneurysm
* Patient's anatomy must be fit for stent graft placement on preoperative angio CT scan.
* Patient is affiliated to the social security or equivalent system.
* The patient must be available for the appropriate follow-up times for the duration of the study.
* Patient has been informed of the nature of the study, agrees to its provisions and has signed the informed consent from.

Exclusion Criteria:

* Patients who do not meet the instructions for use
* Patients with one of the contraindications as indicated in the instructions for use
* Patients with a stenotic internal iliac ostium of < 4mm in Diameter
* Patients with severe internal iliac atherosclerosis
* Patients that do not have a suitable landing area in the main stem of the IIA (maximum diameter in landing area <12mm)
* Patients with pseudoaneurysms
* Patients with symptomatic and ruptured iliac aneurysms
* Patients pretreated with a AAA stent graft or a bifurcated vascular graft
* Patient with thrombocytopenia
* Patient with an estimated glomerular filtration rate < 30 ml/min/1,73m2 immediately before the Intervention
* Female of child bearing potential
* In the lnvestigator's opinion patient has (a) eo-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements, or impact the scientific integrity of the study
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints
* Patient with malignancy needing chemotherapy or radiation
* Patients with life expectancy of less than 36 months
* Patient minor or under guardianship

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with unilateral or bilateral common iliac aneurysm, treated with the E-liac Stent Graft System
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-07 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 30 days follow-up
  Clinical success related to the E-liac Stent Graft combines the following criteria (adapted from Chaikof 2002):
  * Clinical success should be reported on an intent-to-treat Basis
  * requires successful deployment of the E-liac Stent Graft at the intended location without
  * Death as a result of iliac aneurysm-related treatment
  * Type I or III endoleak
  * E-liac Stent Graft infection
  * E-liac Stent Graft thrombosis (including internal iliac artery thrombosis)
  * Aneurysm growth >3mm in maximum diameter for common iliac aneurysm and >5mm in maximum diameter for aortic aneurysm at 12, 24, and 36 months follow-up
  * Common iliac aneurysm rupture
  * Conversion to open repair
  * Failure of E-liac Stent Graft integrity

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Kaladji, Prof., Principal Investigator — CHU Rennes
Locations (2):
- France (2):
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided